CLINICAL TRIAL: NCT04118920
Title: Safety of Topical Insulin Eye Drops for the Treatment of Open-angle Glaucoma
Brief Title: Safety of Topical Insulin Drops for Open-angle Glaucoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE19.154
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma
Keywords: Topical insulin; Dendrite regeneration
MeSH Terms: conditions — Glaucoma | interventions — Insulin; Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: Single-arm prospective open-label interventional study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical insulin (Experimental): Patients will receive topical insulin eye drops.
  Interventions: Drug: Topical insulin (4 units); Drug: Topical insulin (20 units)
- Topical artificial tears (Sham Comparator): Patients will receive topical artificial tears.
  Interventions: Drug: Artificial tears

INTERVENTIONS:
Drug: Topical insulin (4 units) — N=6: 100 U/ml; 4 units of insulin per application; 40 microliters per drop
  Other Names: Humulin R (100 units/mL)
  Arms: Topical insulin
Drug: Topical insulin (20 units) — N=6: 500 U/ml; 20 units of insulin per application; 40 microliters per drop
  Other Names: Entuzity (500 units/mL)
  Arms: Topical insulin
Drug: Artificial tears — N=3, 40 microliters per drop
  Other Names: Refresh Plus Artificial Tears
  Arms: Topical artificial tears

SUMMARY:
Glaucoma, a leading cause of irreversible blindness worldwide, is characterized by a permanent loss of retinal ganglion cells (RGCs), a group of central nervous system (CNS) neurons that convey visual information from the retina to the brain via their long axons. Clinically, axonal damage in RGC results in a loss of visual field and may lead to blindness. Currently, reducing eye pressure remains the sole target of proven glaucoma therapies. However, many patients continue to lose vision even when standard interventions are implemented, accentuating the unmet need for novel therapies.

Dendrites are processes that determine how neurons receive and integrate information. Dendrite retraction and synapse breakdown are early signs of several neurodegenerative disorders. In mammals, CNS neurons have an extremely limited capacity to regenerate after injury. To date, the ability of mammalian neurons to regrow dendrites and reestablish functional synapses has been largely ignored.

Insufficient insulin signaling has been implicated in diseases characterized by dendritic pathology, notably Alzheimer's disease and glaucoma. A versatile hormone, insulin readily crosses the blood-brain-barrier and influences numerous brain processes. In a mouse model of optic nerve transection, our team showed that insulin administration after optic nerve injury promoted robust dendritic regrowth, RGCs survival and retinal responses rescue, providing the first evidence of successful dendrite regeneration in mammalian neurons. Our research validates insulin as a powerful medication to restore dendritic function in glaucoma, forming the basis for using insulin as glaucoma treatment in humans.

Currently, insulin is approved for diabetes. Adverse events of systemic insulin include hypoglycemia, hypokalemia, lipodystrophy, allergies, weight gain, peripheral edema and drug interactions. Experimental use of ocular topical insulin have been tested in small cohorts of healthy individuals and diabetic patients, reporting no significant adverse events. However, these protocols varied in insulin posology and adverse events were only touched upon briefly, indicating the necessity to better characterize the safety profile of such off-label use of insulin before its application as a neuroprotective and regenerative treatment for glaucoma.

In this study, the investigators hypothesize that topical ocular insulin (up to 500 U/ml) at once per day dosing is safe in patients with open angle glaucoma.

DETAILED DESCRIPTION:
Glaucoma: a major health care challenge of the 21st century

Glaucoma is a leading cause of irreversible blindness worldwide and is expected to affect 76 million people by the year 2020. In glaucoma, there is a permanent loss of retinal ganglion cells (RGCs), the long-projecting central nervous system (CNS) neurons that convey visual information from the retina to the brain via their axons. Clinically, such changes translate into a progressive damage of visual field and sometimes result in a complete loss of vision. Currently, intraocular pressure (IOP) reduction remains the sole target of proven glaucoma therapies, consisting of a wide range of eye drops, systemic medications, laser procedures and incisional surgeries. However, many patients continue to lose vision even when these therapies are implemented, exemplifying the unmet need for novel therapies that sustain RGC survival and stimulate their regeneration.

Dendrite pathology: an early sign of neuronal damage in glaucoma Dendrites are specialized processes that determine how neurons receive and integrate information within neuronal circuits. Dendrite retraction and synapse disassembly are early signs of pathology in several psychiatric and neurodegenerative disorders. Dendritic pathology occurs prior to soma or axon loss and correlates with substantial functional deficits. In mammals, CNS neurons have a limited capacity to regenerate after injury. While a large number of studies have focused on axonal regeneration, the ability of mammalian neurons to regrow dendrites and reestablish functional synapses has been largely ignored. This is a critical issue because pathological disconnection from pre-synaptic targets leads to persistent functional impairment and accrued neuronal death, contributing to vision loss in glaucoma.

The role of insulin in dendrite regeneration Aberrant or insufficient insulin signaling, even in the absence of diabetes, has been associated with neurodegeneration in diseases characterized by dendritic pathology, notably Alzheimer's and Parkinson's disease, as well as glaucoma. Traditionally viewed solely as a peripherally acting hormone, insulin crosses the blood-brain-barrier readily and can influence a number of physiological brain processes including neuronal survival, neurotransmission, and cognitive performance. Using a model of optic nerve transection (axotomy), members of our team (Agostinone et al. Brain 2018) showed that insulin administered as eye drops or systemically after dendrites had retracted, promoted robust dendritic growth that restored arbor area and complexity. Remarkably, insulin rescued excitatory postsynaptic sites and light-triggered retinal responses while promoting robust cell survival. This study provides the first evidence of successful dendrite regeneration in mammalian neurons. Unpublished data (manuscript in preparation) from a mouse glaucoma model by our colleagues at the CHUM (Agostinone et al., in preparation) also showed that insulin stimulates similar dendrite regeneration after ocular hypertension damage. These results confirm that injured murine RGCs can effectively regenerate dendrites and validate insulin as a powerful strategy to restore dendritic morphology in glaucoma, providing the basis for need of further investigation of insulin use as glaucoma treatment in humans.

Currently, insulin is approved for subcutaneous or intravenous use as a treatment for diabetes mellitus. Adverse events of systemic insulin include hypoglycemia, hypokalemia,allergies, weight gain, peripheral edema and drug interactions. Experimental use of ocular topical insulin have been tested in small cohorts of healthy individuals and diabetic patients, reporting no significant adverse events. However, these protocols varied in insulin posology and adverse events were only mentioned briefly, if at all, in most of these studies, indicating the necessity of better characterizing the safety profile of such off-label use of insulin prior to implementing its use as neuroprotective and regenerative treatment for glaucoma.

Experimental nature of the medication / treatment:

Topical application of insulin with concentrations of 100 U/ml (Humulin R U-100, Eli Lilly Canada, St-Laurent, Quebec, Canada) and 500 U/ml (Entuzity, Eli Lilly Canada, St-Laurent, Quebec, Canada) once per day to eyes diagnosed with open angle glaucoma. Both products of insulin are approved by Health Canada for subcutaneous and intravenous use for the treatment of diabetes mellitus. The proposed route of administration and indication of insulin use in this current study are therefore of off-label nature, for which the investigators will request a non-objection letter from Health Canada.

Hypothesis of the study: Topical ocular insulin (up to 500 U/ml) at once per day dosing is safe in patients with open angle glaucoma.

Objectives: To document and to report any ocular and/or systemic adverse events associated with topical insulin eye drops.

ELIGIBILITY:
* Please note that this study is only open to patients who are Quebec residents and who are already followed at the Centre Hospitalier de l'Université de Montréal (CHUM).

Inclusion Criteria:

* Age 18-75 years
* Capable to provide informed consent
* Diagnosed of moderate primary open-angle glaucoma
* Moderate glaucoma is defined as:

  * Vertical cup-to-disc ratio of 0.7-0.85 and (or)
  * Moderate VF defect not within 10° of fixation (e.g. mean deviation (MD) from -6 to -12 dB on Humphrey Visual Field 24-2)
* Only one eye per patient will be selected as the study eye - if both eyes meet the inclusion criteria, the eye with the worse acuity and/or visual field will be selected. The contralateral eye will be left untouched.
* Patients with non-restrictive diets (see exclusion criteria for a list of diets considered restrictive).
* Normal serum potassium level (3.5-5.0mEq/L or 3.5-5.0 mMol/L) and HbA1C (≤5.7%) at baseline.

Exclusion Criteria:

* Younger than 18 years of age or older than 75 years of age
* Pregnant or breastfeeding woman
* Presence of any ocular pathologies other than glaucoma that contributes to the severe vision loss (retinopathy/maculopathy, non-glaucomatous optic neuropathy, severe uveitis, keratopathy, etc.)
* History of cataract surgery (complicated or uncomplicated) within 3 months of the study
* Any other intraocular surgery within 6 months of the initiation of the study
* Visual acuity of no light perception (NLP)
* Unable to provide informed consent
* Unable to complete the tests and follow-ups required by the study
* Diagnosis of glucose intolerance, type 1 or 2 diabetes mellitus (HbA1C > 5.7%26)
* Diagnosis of conditions leading to baseline increased risk of hypokalemia and hypoglycemia such as:
* Chronic kidney disease (with or without dialysis)
* Cardiovascular disease, history of arrythmias
* Cirrhosis or other inflammatory liver diseases (hepatitis B and C)
* Inflammatory bowel disease
* Active or chronic infections causing potassium wasting: HIV, tuberculosis, hepatitis, and sepsis as a result of these infections
* Metabolic disorders predisposing to hypokalemia such as: renal tubular acidosis, primary hyperaldosteronism, Cushing's disease
* Potomania or other alcohol abuse
* Hyperhidrosis
* Polyuria
* Nephropathies such as tubulointerstitial diseases or tubular injuries causing salt-wasting
* Any hematologic or inflammatory conditions requiring plasmapheresis
* Any known insulin-secreting tumors
* Patients with restrictive diets
* Patients at risk of malnutrition due to disability limiting daily dietary intake of nutrients and electrolytes ("tea-and-toast diet")
* Veganism
* Medically recommended low-potassium diet (such as chronic kidney disease)
* Eating disorders with risks of malnutrition, such as anorexia nervosa and bulimia
* Use of medications predisposing a patient to the risk of hypokalemia such as high dose diuretics and laxatives
* History of hypersensitivity to insulin or any of the ingredients in the formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of hypoglycemia | 6 months
  Monitor blood glucose levels in patients
Rate of hypokalemia | 6 months
  Monitor serum potassium levels in patients
Rates of other reported adverse events | 6 months
  Monitor any adverse event in patients
Ocular tolerability of the instilled drops | 6 months
  Monitor the ocular tolerability of insulin drops on patients with a visual analog scale of ocular tolerability

SECONDARY OUTCOMES:
Snellen chart visual acuity expressed in logMAR | 6 months
  Monitor visual acuity in patients
Intraocular pressure (IOP) | 6 months
  Monitor IOP in patients
Average retinal nerve fiber layer (RNFL) and ganglion cell complex (GCC) thickness on spectral domain optical coherence tomography (SD-OCT) | 6 months
  Monitor RNFL and GCC thickness in patients
Perfusion density (PD) on optical coherence tomography-angiography (OCT-A) | 6 months
  Monitor PD on OCT-A
Flow index (FI) on OCT-A | 6 months
  Monitor FI on OCT-A
Visual field index (VFI) on Swedish Interactive Thresholding Algorithm (SITA) 24-2 visual field | 6 months
  Monitor VFI on patients' visual fields
Mean deviation (MD) and pattern standard deviation (PSD) on SITA 24-2 visual field | 6 months
  Monitor MD and PSD on patients' visual fields

CONTACTS AND LOCATIONS:
Overall Officials: Qianqian Wang, MD, FRCSC, Principal Investigator — Département d'ophtalmologie, Centre hospitalier de l'Université de Montréal
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940
- [Background] Agostinone J, Di Polo A. Retinal ganglion cell dendrite pathology and synapse loss: Implications for glaucoma. Prog Brain Res. 2015;220:199-216. doi: 10.1016/bs.pbr.2015.04.012. Epub 2015 Jun 30. PMID 26497792
- [Background] Canadian Ophthalmological Society Glaucoma Clinical Practice Guideline Expert Committee; Canadian Ophthalmological Society. Canadian Ophthalmological Society evidence-based clinical practice guidelines for the management of glaucoma in the adult eye. Can J Ophthalmol. 2009;44 Suppl 1:S7-93. doi: 10.3129/cjo44s1. No abstract available. English, French. PMID 19492005
- [Background] Schwartz M, London A. Glaucoma as a neuropathy amenable to neuroprotection and immune manipulation. Prog Brain Res. 2008;173:375-84. doi: 10.1016/S0079-6123(08)01126-6. PMID 18929122
- [Background] Frankfort BJ, Khan AK, Tse DY, Chung I, Pang JJ, Yang Z, Gross RL, Wu SM. Elevated intraocular pressure causes inner retinal dysfunction before cell loss in a mouse model of experimental glaucoma. Invest Ophthalmol Vis Sci. 2013 Jan 28;54(1):762-70. doi: 10.1167/iovs.12-10581. PMID 23221072
- [Background] Pang JJ, Frankfort BJ, Gross RL, Wu SM. Elevated intraocular pressure decreases response sensitivity of inner retinal neurons in experimental glaucoma mice. Proc Natl Acad Sci U S A. 2015 Feb 24;112(8):2593-8. doi: 10.1073/pnas.1419921112. Epub 2015 Feb 9. PMID 25675503
- [Background] Hilliard MA. Axonal degeneration and regeneration: a mechanistic tug-of-war. J Neurochem. 2009 Jan;108(1):23-32. doi: 10.1111/j.1471-4159.2008.05754.x. Epub 2008 Nov 15. PMID 19054282
- [Background] Kleinridders A. Deciphering Brain Insulin Receptor and Insulin-Like Growth Factor 1 Receptor Signalling. J Neuroendocrinol. 2016 Nov;28(11):10.1111/jne.12433. doi: 10.1111/jne.12433. PMID 27631195
- [Background] Ghasemi R, Haeri A, Dargahi L, Mohamed Z, Ahmadiani A. Insulin in the brain: sources, localization and functions. Mol Neurobiol. 2013 Feb;47(1):145-71. doi: 10.1007/s12035-012-8339-9. Epub 2012 Sep 7. PMID 22956272
- [Background] Agostinone J, Alarcon-Martinez L, Gamlin C, Yu WQ, Wong ROL, Di Polo A. Insulin signalling promotes dendrite and synapse regeneration and restores circuit function after axonal injury. Brain. 2018 Jul 1;141(7):1963-1980. doi: 10.1093/brain/awy142. PMID 29931057
- [Background] Bartlett JD, Turner-Henson A, Atchison JA, Woolley TW, Pillion DJ. Insulin administration to the eyes of normoglycemic human volunteers. J Ocul Pharmacol. 1994 Winter;10(4):683-90. doi: 10.1089/jop.1994.10.683. PMID 7714412
- [Background] Bartlett JD, Slusser TG, Turner-Henson A, Singh KP, Atchison JA, Pillion DJ. Toxicity of insulin administered chronically to human eye in vivo. J Ocul Pharmacol. 1994 Spring;10(1):101-7. doi: 10.1089/jop.1994.10.101. PMID 8207318
- [Background] Wang AL, Weinlander E, Metcalf BM, Barney NP, Gamm DM, Nehls SM, Struck MC. Use of Topical Insulin to Treat Refractory Neurotrophic Corneal Ulcers. Cornea. 2017 Nov;36(11):1426-1428. doi: 10.1097/ICO.0000000000001297. PMID 28742619
- [Background] Fai S, Ahem A, Mustapha M, Mohd Noh UK, Bastion MC. Randomized Controlled Trial of Topical Insulin for Healing Corneal Epithelial Defects Induced During Vitreoretinal Surgery in Diabetics. Asia Pac J Ophthalmol (Phila). 2017 Sep-Oct;6(5):418-424. doi: 10.22608/APO.201780. Epub 2017 Aug 22. PMID 28828764
- [Background] Bastion ML, Ling KP. Topical insulin for healing of diabetic epithelial defects?: A retrospective review of corneal debridement during vitreoretinal surgery in Malaysian patients. Med J Malaysia. 2013 Jun;68(3):208-16. PMID 23749008
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S64-71. doi: 10.2337/dc12-s064. No abstract available. PMID 22187472
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Background] SA J. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics. 2005;4(4):287-91.
- [Background] Information for the Physician: Humulin R Regular Insulin Human Injection, USP, (rDNA origin) 100 units per ml (U-100). In: Administration FaD, editor.: Lilly USA; 2011.